CLINICAL TRIAL: NCT00242736
Title: An Open-Label Study of Once-Daily Oral Administration of Esomeprazole 40 mg in Patients With Symptoms of Gastroesophageal Reflux Disease (GERD) to Investigate the Relationship Between the Presence of Erosive Esophagitis (EE) at Baseline and Heartburn Resolution After 4 Weeks of Treatment
Brief Title: An Open-Label Study of Once-Daily Oral Administration of Esomeprazole 40 mg in Patients With Symptoms of Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00083
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
The purpose of this study is to evaluate whether there is a difference in proportion of patients with resolution of heartburn and other symptoms related to gastroesophageal reflux disease (GERD) after four weeks of treatment with esomeprazole (NEXIUM®) in those subjects with Erosive Esophagitis (EE) and those without EE.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of GERD as defined in this protocol: Heartburn (severity of mild, moderate or severe) 2 or more times in the 7 days prior to the Screening visit (Visit 1) and, on average, at least 2 times per week over the past 3 months.
* Male or female, 18 to 70 years old, inclusive.
* Non-pregnant, non-lactating female patients. Female patients must be postmenopausal, surgically sterile, or using a medically acceptable form of birth control, as determined by the investigator. Females of childbearing potential must agree to continue using an acceptable form of birth control throughout the conduct of the study.
* Negative urine pregnancy test for females of childbearing potential.
* Willingness to adhere to all protocol requirements.

Exclusion Criteria:

* Previous enrollment in the present study.
* Significant clinical illness within 2 weeks prior to the first dose of study medication or a significant illness during the study.
* Use of a PPI, including PRILOSEC OTC®, within 21 days of Screening (Visit 1) or at anytime during the study (Visit 1 through Visit 4).
* Daily therapy with an H2 RA within 14 days of Screening (Visit 1): eg, ranitidine (ZANTAC®), cimetidine (TAGAMET®), nizatidine (AXID®), famotidine (PEPCID®) (occasional use; ie, less than daily, is permitted).
* Use of H2 RAs at any frequency are prohibited throughout the entire study (Visit 1 through Visit 4).
* A history of gastric or esophageal surgery (including, but not limited to, Nissen fundoplication and bariatric surgery), except for simple closure of a perforated ulcer or procedures that would not affect the study as determined by the Clinical Study Team physician at AstraZeneca.
* Clinically significant gastrointestinal (GI) bleeding (eg, melena, frank hematochezia) within 3 days of Screening (Visit 1) or noted at the time of baseline EGD.
* Non-acid related etiologies of esophagitis (eg, pill-induced, caustic ingestion or eosinophilic esophagitis).

Generalized bleeding disorders resulting from hemorrhagic diathesis (such as abnormalities in clotting factors or platelets).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2005-10; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
The outcome variable will be the percentage of patients with heartburn resolution stratified by the presence or absence of EE

SECONDARY OUTCOMES:
The outcome variables will be resolution of acid regurgitation, dysphagia, and epigastric pain symptoms after 2 and 4 weeks of treatment.
The outcome variable will be the resolution of heartburn after 2 weeks of treatment.
The outcome variables will be the presence or absence of EE at baseline and the resolution of heartburn at the end of the 4-week treatment period.
The outcome variable used for this objective will be the percentage of endoscoped patients with EE (LA Classification Grades A-D) at baseline.
Safety variables that will be measured and tabulated include adverse events, laboratory evaluations, physical exams, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (25):
- United States (25):
  - Research Site, Alabaster, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, North Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Orange, California
  - Research Site, Torrance, California
  - Research Site, Miami, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Arlington Heights, Illinois
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Hollywood, Maryland
  - Research Site, Elkin, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Christiansburg, Virginia
  - Research Site, Norfolk, Virginia

REFERENCES:
- [Derived] Orlando RC, Monyak JT, Silberg DG. Predictors of heartburn resolution and erosive esophagitis in patients with GERD. Curr Med Res Opin. 2009 Sep;25(9):2091-102. doi: 10.1185/03007990903080931. PMID 19601705